CLINICAL TRIAL: NCT04398940
Title: A Single-arm, Multicenter Study to Evaluate the Efficacy and Safety of TQ-B3139 in Subjects With MET-Altered Advanced Non-small Cell Lung Cancer
Brief Title: A Study of TQ-B3139 Capsules in Subjects With MET-Altered Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3139-II-02
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2019-11

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3139 capsules (Experimental): TQ-B3139 capsules administered orally.
  Interventions: Drug: TQ-B3139

INTERVENTIONS:
Drug: TQ-B3139 — TQ-B3139 capsules administered 600mg orally, twice daily in 28-day cycle.

SUMMARY:
This is a single-arm, multi-center clinical trial to evaluate the safety and efficacy of TQ-B3139 capsules in patients with MET gene abnormal advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1; 2. Life expectancy ≥12 weeks; 3. MET-altered non-small cell lung cancer (NSCLC) ; 4. Has at least one measurable lesion; 5. Previous standard treatment has failed; 6. Adequate organ system function; 7. Left ventricular ejection fraction (LVEF) ≥50%; 8. Understood and signed an informed consent form.

Exclusion Criteria:

* 1. Has diagnosed and/or treated additional malignancy within 3 years prior to the first administration; 2. Has received c-MET inhibitors; 3. Has received other system anti-tumor treatment within 4 weeks before the first administration; 4. Has received major surgical treatment within 4 weeks before the first administration; 5. Has received radiotherapy or any surgery within 2 weeks before the first administration; 6. Acute toxicity that is ≥ Grade 2 caused by previous cancer therapy; 7. Has active infection within 2 weeks before the first administration; 8. Has currently uncontrollable congestive heart failure; 9. Has currently uncontrollable congestive heart failure; 10. Has continuous arrhythmia ≥ Grade 2, uncontrollable atrial fibrillation or QTc interval > 480ms; 11. Has uncontrollable effusion; 12. Has interstitial lung diseases; 13. Has severely unstable central nervous system metastasis; 14. Has active viral infection; 15. Has multiple factors affecting oral medication; 16. Breastfeeding or pregnant women; Men unwilling to use adequate contraceptive measures during the study; 17. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 18 months
  Percentage of subjects achieving complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 18 months
  PFS was defined as the time from the date of study enrollment to the date of the first of the following events, objective disease progression or death due to any cause.
Disease control rate (DCR) | up to 18 months
  Percentage of subjects achieving complete response (CR) and partial response (PR) and stable disease (SD).
Overall survival (OS) | up to 24 months
  OS defined as the time from the first dose to death from any cause. Survival time was censored at the date of last contact for patients who were still alive or lost to follow-up.
Duration of Response (DOR) | up to 18 months
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.
Intracranial progression-free survival (CNS-PFS) | up to 18 months
  The time from enrollment to the first confirmed intracranial progression for brain metastases.
Intracranial objective response rate (CNS-ORR) | up to 18 months
  Percentage of subjects achieving intracranial complete response and partial response.
Time to progress of intracranial disease (CNS-TTP) | up to 18 months
  The time from the first dose to the first occurrence of intracranial disease progression.

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Sixth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Sir Run Shaw Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality